CLINICAL TRIAL: NCT00614120
Title: Effect of Liraglutide or Glimepiride Added to Metformin on Glycaemic Control in Subjects With Type 2 Diabetes
Brief Title: Effect of Liraglutide or Glimepiride Added to Metformin on Blood Glucose Control in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1796
Record Dates: First submitted 2008-01-15; First posted 2008-02-13 (Estimated); Results first posted 2010-03-12 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; glimepiride; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lira 0.6 + Met (Experimental): Liraglutide 0.6 mg + metformin + glimepiride placebo
  Interventions: Drug: liraglutide; Drug: placebo; Drug: metformin
- Lira 1.2 + Met (Experimental): Liraglutide 1.2 mg + metformin + glimepiride placebo
  Interventions: Drug: placebo; Drug: liraglutide; Drug: metformin
- Lira 1.8 + Met (Experimental): Liraglutide + metformin + glimepiride placebo
  Interventions: Drug: placebo; Drug: liraglutide; Drug: metformin
- Glim + Met (Experimental): Glimepiride 4.0 mg + metformin + liraglutide placebo
  Interventions: Drug: glimepiride; Drug: metformin; Drug: placebo

INTERVENTIONS:
Drug: liraglutide — 0.6 mg/day, s.c. (under the skin) injection
  Arms: Lira 0.6 + Met
Drug: placebo — Glimepiride placebo, capsules
  Arms: Lira 0.6 + Met; Lira 1.2 + Met; Lira 1.8 + Met
Drug: liraglutide — 1.2 mg/day, s.c. (under the skin) injection
  Arms: Lira 1.2 + Met
Drug: liraglutide — 1.8 mg/day, s.c. (under the skin) injection
  Arms: Lira 1.8 + Met
Drug: glimepiride — Capsules, 4.0 mg/day
  Arms: Glim + Met
Drug: metformin — Tablets, 1.5-2.0 g/day
Drug: placebo — Liraglutide placebo, s.c. (under the skin) injection
  Arms: Glim + Met

SUMMARY:
This trial is conducted in Asia. The trial is designed to compare the effect on glycaemic control of liraglutide or glimepiride added to metformin in subjects with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Subjects diagnosed with type 2 diabetes and treated with one or more oral antidiabetic drugs (OADs) for the last 3 months
* HbA1c: 7.0-11.0% (both incl.) for subjects on OAD alone
* HbA1c: 7.0-10.0 % (both incl.) for subjects on OAD combination therapy
* BMI less than 45.0 kg/m^2

Exclusion Criteria:

* Treatment with insulin within the last 3 months prior to the trial
* Impaired liver or/and renal function
* Significant cardiovascular disease over the last 6 months
* Known retinopathy or maculopathy
* Recurrent major hypoglycaemia or hypoglycaemic unawareness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 929 (Actual)
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), MD, PhD, Study Director — Novo Nordisk A/S
Locations (41):
- China (14):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Chongqing, Chongqing Municipality
  - Novo Nordisk Investigational Site, Fuzhou, Fujian
  - Novo Nordisk Investigational Site, Harbin, Heilongjiang
  - Novo Nordisk Investigational Site, Wuhan, Hubei
  - Novo Nordisk Investigational Site, Nanjing, Jiangsu
  - Novo Nordisk Investigational Site, Suzhou, Jiangsu
  - Novo Nordisk Investigational Site, Wuxi, Jiangsu
  - Novo Nordisk Investigational Site, Xi'an, Shaanxi
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
  - Novo Nordisk Investigational Site, Hangzhou, Zhejiang
  - Novo Nordisk Investigational Site, Shenyang
  - Novo Nordisk Investigational Site, Tianjin
  - Novo Nordisk Investigational Site, Wuhan
- India (22):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Hyderbad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Kochi, Kerala
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Bhubaneswar, Odisha
  - Novo Nordisk Investigational Site, Jaipur, Rajasthan
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Madurai, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Ghaziabad
  - Novo Nordisk Investigational Site, Kochi
  - Novo Nordisk Investigational Site, Kolkata
  - Novo Nordisk Investigational Site, Mumbai
  - Novo Nordisk Investigational Site, New Delhi
  - Novo Nordisk Investigational Site, Patna
  - Novo Nordisk Investigational Site, Secunderabad
  - Novo Nordisk Investigational Site, Trivandrum
  - Novo Nordisk Investigational Site, Visakhapatnam
- South Korea (5):
  - Novo Nordisk Investigational Site, Goyang
  - Novo Nordisk Investigational Site, Incheon
  - Novo Nordisk Investigational Site, Seoul
  - Novo Nordisk Investigational Site, Sungnam
  - Novo Nordisk Investigational Site, Suwon

REFERENCES:
- [Result] Yang W, Chen L, Ji Q, Liu X, Ma J, Tandon N, Bhattacharyya A, Kumar A, Kim KW, Yoon KH, Bech OM, Zychma M. Liraglutide provides similar glycaemic control as glimepiride (both in combination with metformin) and reduces body weight and systolic blood pressure in Asian population with type 2 diabetes from China, South Korea and India: a 16-week, randomized, double-blind, active control trial(*). Diabetes Obes Metab. 2011 Jan;13(1):81-8. doi: 10.1111/j.1463-1326.2010.01323.x. PMID 21114607
- [Result] Alves C, Batel-Marques F, Macedo AF. A meta-analysis of serious adverse events reported with exenatide and liraglutide: acute pancreatitis and cancer. Diabetes Res Clin Pract. 2012 Nov;98(2):271-84. doi: 10.1016/j.diabres.2012.09.008. Epub 2012 Sep 23. PMID 23010561
- [Result] Jensen TM, Saha K, Steinberg WM. Is there a link between liraglutide and pancreatitis? A post hoc review of pooled and patient-level data from completed liraglutide type 2 diabetes clinical trials. Diabetes Care. 2015 Jun;38(6):1058-66. doi: 10.2337/dc13-1210. Epub 2014 Dec 12. PMID 25504028
- [Result] Ingwersen SH, Petri KC, Tandon N, Yoon KH, Chen L, Vora J, Yang W. Liraglutide pharmacokinetics and dose-exposure response in Asian subjects with Type 2 diabetes from China, India and South Korea. Diabetes Res Clin Pract. 2015 Apr;108(1):113-9. doi: 10.1016/j.diabres.2015.01.001. Epub 2015 Jan 19. PMID 25684604
- [Derived] Buse JB, Garber A, Rosenstock J, Schmidt WE, Brett JH, Videbaek N, Holst J, Nauck M. Liraglutide treatment is associated with a low frequency and magnitude of antibody formation with no apparent impact on glycemic response or increased frequency of adverse events: results from the Liraglutide Effect and Action in Diabetes (LEAD) trials. J Clin Endocrinol Metab. 2011 Jun;96(6):1695-702. doi: 10.1210/jc.2010-2822. Epub 2011 Mar 30. PMID 21450987
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 51 centres in three countries: China (17), India (24) and South Korea (10)
Pre-assignment Details: A metformin run-in period of 3 weeks followed by a metformin maintenance period of 3 weeks before randomisation with dose levels increased to 2000 mg/day. Subjects already on metformin therapy at enrolment could go through a modified titration period or advance directly to the metformin maintenance period at the discretion of the investigator.
Groups:
- Lira 0.6 + Met: Liraglutide 0.6 mg once daily + metformin 1.5-2.0 g daily + glimepiride placebo
- Lira 1.2 + Met: Liraglutide 1.2 mg once daily + metformin 1.5-2.0 g daily + glimepiride placebo
- Lira 1.8 + Met: Liraglutide 1.8 mg once daily + metformin 1.5-2.0 g daily + glimepiride placebo
- Glim + Met: Glimepiride 4.0 mg + metformin 1.5-2.0 g daily + liraglutide placebo
Period: Overall Study
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Glim + Met
Started | 231 (Randomised) | 233 (Randomised) | 234 (Randomised) | 231 (Randomised)
Exposed to Study Drug | 231 | 233 | 233 (Subject withdrew before exposure to study products, and thus not included in full analysis set.) | 231
Completed | 202 | 187 | 175 | 215
Not Completed | 29 | 46 | 59 | 16
Not completed — Adverse Event | 9 | 22 | 30 | 3
Not completed — Lack of Efficacy | 3 | 3 | 2 | 2
Not completed — Protocol Violation | 2 | 5 | 3 | 1
Not completed — Withdrawal criteria | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 10 | 16 | 3
Not completed — Did not meet trial criteria | 0 | 1 | 1 | 1
Not completed — hCG positive (not pregnant) | 0 | 0 | 1 | 0
Not completed — Hypoglycaemia | 0 | 0 | 0 | 1
Not completed — Lack of trial product | 3 | 3 | 2 | 0
Not completed — Late syphilis, latent | 1 | 0 | 0 | 0
Not completed — Taken inhibition medication eg Prandin | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 1 | 2 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Glim + Met | Total
Number analyzed (Participants) | 231 | 233 | 234 | 231 | 929
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (9.5) | 53.5 (9.6) | 52.7 (9.1) | 53.6 (9.7) | 53.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 105 | 108 | 96 | 415
  Male | 125 | 128 | 126 | 135 | 514
Previous OAD treatment [Number; unit: participants] — OAD = Oral Anti-Diabetic Drug
  participants
    Mono-therapy | 72 | 74 | 75 | 68 | 289
    Combination therapy | 159 | 159 | 159 | 163 | 640
BMI [Mean (Standard Deviation); unit: kg/m2] — Body Mass Index
  kg/m2 | 25.9 (4.2) | 25.4 (3.7) | 25.8 (3.8) | 25.3 (3.7) | 25.6 (3.8)
Duration of diabetes [Mean (Standard Deviation); unit: years] — Number of years since diagnosis
  years | 7.4 (5.4) | 7.5 (5.3) | 7.2 (5.2) | 7.8 (6.1) | 7.5 (5.5)
Height [Mean (Standard Deviation); unit: m] | 1.63 (0.09) | 1.63 (0.09) | 1.62 (0.08) | 1.64 (0.09) | 1.63 (0.09)
Weight [Mean (Standard Deviation); unit: kg] | 68.6 (11.6) | 67.4 (11.3) | 68.2 (11.9) | 68.2 (11.9) | 68.1 (11.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin A1c (HbA1c)
Description: Percentage point change in Glycosylated Haemoglobin A1c (HbA1c) from baseline (week 0) to 16 weeks (end of treatment).
Time Frame: week 0, week 16
Population: The Full Analysis Set (FAS) using LOCF (Last Observation Carried Forward) is all randomised subjects who had been exposed to at least one dose of the study products.
Measure: Mean (Standard Deviation); unit: percentage point of total HbA1c
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Glim + Met
Number analyzed (Participants) | 226 | 222 | 221 | 230
percentage point of total HbA1c | -1.0 (1.04) | -1.3 (1.09) | -1.4 (1.23) | -1.3 (0.98)
Statistical Analysis 1: Comparison: Lira 1.8 + Met vs Glim + Met; Based on standard normal theory, the sample size needed in order to be able to show that lira + met is non-inferior to glim + met when using a 1:1 randomisation and a non-inferiority criteria of 0.4% with a power of at least 85%, is tabulated below using different SD of HbA1c. Assuming a drop out rate of 25%, the total number of subjects to be randomised is 896 (224 for each dose of the liraglutide + metformin group and 224 subjects in metformin+glimepiride treatment group) with a SD of 1.2%; Test type: Non-Inferiority or Equivalence — Non-inferiority is concluded if the two-sided upper limit of the 95% confidence interval for treatment difference in mean change in HbA1c between lira 1.8mg + met and glim + met is below 0.4%; p < 0.0001, ANCOVA — Non-inferiority; <.0001. In order to protect the overall Type I error rate when testing for non-inferiority of the three doses of lira + met to glim + met, the comparisons will be invoked sequentially for descending doses of liraglutide; ANCOVA model with treatment, country and previous treatment as fixed effects and baseline value as a covariate; Estimated treatment difference, LS Mean = -0.06, 95% CI [-0.23 to 0.11] — The p-values correspond to one-sided hypotheses of either superiority or non-inferiority. Statistical significance on a 2.5% level
Statistical Analysis 2: Comparison: Lira 1.2 + Met vs Glim + Met; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority is concluded if the two-sided upper limit of the 95% confidence interval for treatment difference in mean change in HbA1c between lira 1.2mg + met and glim + met is below 0.4%; p < .0001, ANCOVA — In order to protect the overall Type I error rate when testing for non-inferiority of the three doses of lira + met to glim + met, the comparisons will be invoked sequentially for descending doses of liraglutide; ANCOVA model with treatment, country and previous treatment as fixed effects and baseline value as a covariate; Estimated treatment difference, LS Mean = 0.03, 95% CI [-0.14 to 0.20] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Lira 0.6 + Met vs Glim + Met; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Non-inferiority is concluded if the two-sided upper limit of the 95% confidence interval for treatment difference in mean change in HbA1c between lira 0.6mg + met and glim + met is below 0.4%; p = 0.0421, ANCOVA — [p-value comment as in outcome 1, analysis 2]; ANCOVA model with treatment, country and previous treatment as fixed effects and baseline value as a covariate; Estimated treatment difference, LS Mean = 0.25, 95% CI [0.08 to 0.42] — The p-values correspond to one-sided hypotheses of either superiority or non-inferiority

2. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline (week 0) to 16 weeks (end of treatment)
Time Frame: week 0, week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Glim + Met
Number analyzed (Participants) | 227 | 225 | 224 | 231
kg | -1.8 (2.2) | -2.3 (2.4) | -2.4 (2.6) | 0.1 (2.2)

3. Secondary Outcome: Change in Self-measured Fasting Plasma Glucose
Description: Change in self-measured fasting plasma glucose from baseline (week 0) to 16 weeks (end of treatment). Self-measurement of plasma glucose was performed using a glucose meter and subjects were instructed to record self-measured plasma glucose values into a diary.
Time Frame: week 0, week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Glim + Met
Number analyzed (Participants) | 224 | 226 | 222 | 229
mg/dL | -1.83 (2.66) | -1.96 (2.35) | -2.28 (2.94) | -2.13 (2.25)

4. Secondary Outcome: 7-point Self-measured Plasma Glucose Profiles
Description: Summary of 7-Point Profiles of Self-Measured Plasma Glucose by Treatment, Week and Time. The 7 time points for self-measurements for all treatment groups were: Before each meal (breakfast, lunch and dinner), at 90 min after start of each meal (breakfast, lunch and dinner) and at bedtime, measured over 16 weeks of treatment (at week 0, 8, 12 and 16).
Time Frame: week 0, 8, 12 and 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Glim + Met
Number analyzed (Participants) | 231 | 233 | 233 | 231
mg/dl
  Week 0 - Before breakfast | 168.2 (43.5) | 167.5 (42.5) | 168.8 (40.4) | 163.8 (41.2)
  Week 0 - 90 minutes after breakfast | 245.9 (71.6) | 248.0 (70.0) | 245.4 (63.8) | 238.5 (62.4)
  Week 0 - Before lunch | 178.5 (62.7) | 180.5 (63.5) | 176.9 (56.8) | 175.8 (61.0)
  Week 0 - 90 minutes after lunch | 234.2 (68.7) | 232.3 (67.0) | 234.4 (64.2) | 227.6 (67.0)
  Week 0 - Before dinner | 194.8 (63.0) | 184.8 (65.0) | 190.9 (61.7) | 180.2 (59.2)
  Week 0 - 90 minutes after dinner | 239.6 (65.3) | 239.6 (71.3) | 244.0 (69.8) | 231.6 (60.3)
  Week 0 - Bedtime | 205.7 (69.6) | 208.1 (67.5) | 219.3 (71.7) | 202.7 (66.4)
  Week 8 - Before breakfast | 137.0 (31.2) | 130.4 (28.0) | 133.7 (28.4) | 130.1 (31.8)
  Week 8 - 90 minutes after breakfast | 198.5 (55.8) | 190.1 (50.8) | 178.5 (48.2) | 201.2 (54.4)
  Week 8 - Before lunch | 144.8 (45.2) | 136.5 (41.8) | 138.0 (37.8) | 132.6 (46.1)
  Week 8 - 90 minutes after lunch | 187.2 (48.7) | 176.9 (49.5) | 177.9 (48.4) | 184.3 (54.2)
  Week 8 - Before dinner | 159.1 (47.5) | 147.8 (40.1) | 144.2 (40.6) | 143.3 (47.8)
  Week 8 - 90 minutes after dinner | 193.7 (53.2) | 187.1 (49.3) | 183.3 (53.9) | 190.2 (51.7)
  Week 8 - Bedtime | 169.1 (51.5) | 161.6 (47.1) | 155.8 (45.6) | 163.6 (50.5)
  Week 12 - Before breakfast | 137.8 (33.6) | 130.2 (25.0) | 130.2 (26.8) | 128.5 (29.7)
  Week 12 - 90 minutes after breakfast | 197.5 (54.2) | 185.7 (49.4) | 178.6 (51.6) | 200.8 (57.9)
  Week 12 - Before lunch | 141.8 (48.3) | 135.6 (40.3) | 134.1 (40.3) | 129.3 (47.7)
  Week 12 - 90 minutes after lunch | 183.7 (50.0) | 174.7 (46.2) | 173.7 (53.1) | 185.3 (52.0)
  Week 12 - Before dinner | 156.4 (44.8) | 143.4 (36.1) | 144.5 (43.0) | 144.2 (49.2)
  Week 12 - 90 minutes after dinner | 197.2 (51.8) | 185.7 (47.1) | 183.5 (51.7) | 188.5 (50.1)
  Week 12 - Bedtime | 168.2 (52.1) | 158.9 (45.3) | 158.9 (47.0) | 159.9 (47.6)
  Week 16 - Before breakfast | 137.3 (31.2) | 132.9 (26.4) | 128.6 (26.1) | 131.0 (35.3)
  Week 16 - 90 minutes after breakfast | 195.6 (57.1) | 188.7 (51.6) | 177.6 (51.6) | 195.1 (57.4)
  Week 16 - Before lunch | 140.5 (41.3) | 137.0 (40.3) | 137.8 (40.8) | 128.8 (45.4)
  Week 16 - 90 minutes after lunch | 185.8 (44.4) | 181.4 (46.7) | 173.2 (50.7) | 182.2 (51.8)
  Week 16 - Before dinner | 151.5 (38.5) | 148.4 (39.8) | 140.9 (38.8) | 144.9 (45.3)
  Week 16 - 90 minutes after dinner | 195.0 (52.2) | 183.3 (46.2) | 173.2 (48.3) | 192.6 (53.8)
  Week 16 - Bedtime | 166.4 (50.6) | 159.8 (44.7) | 151.6 (40.3) | 157.7 (47.6)

5. Secondary Outcome: Change in Beta-cell Function
Description: Change in beta cell function from baseline (week 0) to 16 weeks (end of treatment). Beta-cell function was derived from fasting plasma glucose (FPG) and fasting insulin concentrations using the homeostasic model assessment (HOMA) method which uses the assumption that normal-weight normal subjects aged under 35 years have a 100% beta-cell function (HOMA-B).
  Beta-cell function: HOMA-B (%) = 20∙fasting insulin[uU/mL] divided by (FPG mmol/L]-3.5).
Time Frame: week 0, week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage point (%point)
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Glim + Met
Number analyzed (Participants) | 216 | 216 | 213 | 222
percentage point (%point) | 15.3 (94.6) | 17.8 (30.4) | 21.7 (78.5) | 21.8 (43.1)

6. Secondary Outcome: Change in Fasting Lipid Profile
Description: Change in fasting lipid profiles from baseline (week 0) to 16 weeks (end of treatment). Fasting lipid profiles is based on:
  * Total Cholesterol (TC)
  * Low-density Lipoprotein-cholesterol (LDL-C)
  * Very Low-density Lipoprotein-cholesterol (VLDL-C)
  * High-density Lipoprotein-cholesterol (HDL-C)
  * Triglyceride (TG)
  * Free Fatty Acid (FFA)
Time Frame: week 0, week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Glim + Met
Number analyzed (Participants) | 231 | 233 | 233 | 231
mmol/L
  Change in TC (Absolute), N=221, 216, 216, 228 | 0.06 (0.74) | -0.01 (0.77) | -0.03 (0.73) | 0.02 (0.73)
  Change in LDL-C (Absolute), N=221, 216, 216, 228 | 0.06 (0.61) | -0.03 (0.64) | 0.00 (0.58) | 0.04 (0.55)
  Change in VLDL-C (Absolute), N=213, 210, 207, 220 | 0.03 (0.35) | 0.05 (0.40) | 0.01 (0.35) | 0.05 (0.42)
  Change in HDL-C (Absolute), N=217, 212, 212, 220 | -0.02 (0.19) | -0.05 (0.34) | -0.05 (0.15) | -0.01 (0.34)
  Change in TG (Absolute), N=220, 212, 213, 226 | -0.08 (0.96) | -0.06 (1.13) | -0.22 (1.57) | -0.07 (1.26)
  Change in FFA (Absolute), N=218, 214, 216, 227 | -0.03 (0.28) | -0.04 (0.28) | -0.10 (0.28) | -0.02 (0.28)

7. Secondary Outcome: Change in Fasting Lipid Profile, APO-B
Description: Change in fasting lipid profiles based on apolipoprotein B (Apo-B) from baseline (week 0) to 16 weeks (end of treatment).
Time Frame: week 0, week 16
Population: as for outcome 1
Measure: Median (Standard Deviation); unit: g/L
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Glim + Met
Number analyzed (Participants) | 221 | 216 | 216 | 228
g/L | 0.02 (0.17) | 0.00 (0.18) | -0.00 (0.16) | 0.01 (0.17)

8. Secondary Outcome: Hypoglycaemic Episodes
Description: Total number of hypoglycaemic episodes over 16 weeks of treatment occurring from baseline (week 0) to end of treatment (week 16). Hypoglycaemic episodes were defined as major, minor, or symptoms only. Major if the subject was unable to treat her/himself. Minor if subject was able to treat her/himself and plasma glucose was below 3.1 mmol/L. Symptoms only if subject was able to treat her/himself and with no plasma glucose measurement or plasma glucose higher than or equal to 3.1 mmol/L.
Time Frame: weeks 0-16
Population: Safety Analysis Set is all randomised subjects who have been exposed to at least one dose of study products.
Measure: Number; unit: episodes
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Glim + Met
Number analyzed (Participants) | 231 | 233 | 233 | 231
episodes
  Major | 0 | 0 | 0 | 2
  Minor | 6 | 0 | 5 | 80
  Symptoms only | 12 | 11 | 9 | 86

ADVERSE EVENTS:
Time Frame: The adverse events were collected over a time span of 16 weeks.
Description: The safety analysis set is all who had been exposed to at least one dose of the study products.
Arm/Group | Lira 0.6 + Met | Lira 1.2 + Met | Lira 1.8 + Met | Glim + Met
Serious Adverse Events (participants affected / at risk) | 4/231 | 8/233 | 4/233 | 4/231
Other Adverse Events (participants affected / at risk) | 67/231 | 98/233 | 113/233 | 30/231
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira 0.6 + Met (N=231) | Lira 1.2 + Met (N=233) | Lira 1.8 + Met (N=233) | Glim + Met (N=231)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Adams-Stokes syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Brain injury (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cubital tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign hydatidiform mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cryptogenic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira 0.6 + Met (N=231) | Lira 1.2 + Met (N=233) | Lira 1.8 + Met (N=233) | Glim + Met (N=231)
Diarrhoea (Gastrointestinal disorders) | 28 (29) | 36 (43) | 40 (50) | 20 (25)
Nausea (Gastrointestinal disorders) | 29 (33) | 32 (36) | 38 (40) | 5 (5)
Vomiting (Gastrointestinal disorders) | 17 (18) | 22 (22) | 33 (35) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 16 (17) | 12 (13) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 7 (7) | 33 (33) | 35 (35) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 10 (10) | 12 (12) | 7 (7) | 1 (1)
Asthenia (General disorders) | 4 (4) | 10 (10) | 12 (14) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any investigator plans for publication and to review any scientific paper, presentation, communication and other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.